CLINICAL TRIAL: NCT04347434
Title: Assessment of the Effects of Long-term Lipid-lowering Therapy on Parameters of Electrical Myocardial Heterogeneity, Myocardial Deformation Characteristics, Vascular Rigidity, and Quality of Life in Patients With Primary STEMI or NSTEMI
Brief Title: Assessment of the Effects of Long-term Lipid-lowering Therapy in Patients With Primary STEMI or NSTEMI
Acronym: CONTRAST-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Penza State University (Other)
Responsible Party: Principal Investigator, Valentin Oleynikov, DM, Penza State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSU/T-471
Record Dates: First submitted 2020-03-20; First posted 2020-04-15 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction, Acute; Myocardial Strain; Arterial Stiffness; Quality of Life
Keywords: STEMI; NSTEMI; myocardial strain,; arterial stiffness,; lipid-lowering therapy,; electrical myocardial heterogeneity
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Initially, hypolipidemic treatment with atorvastatin at a dose of 80 mg / day is prescribed from the first 24-96 hours of AMI in addition to standard therapy for the disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin 80 mg (Experimental): Treatment with atorvastatin is prescribed at a dose of 80 mg / day from the first 24-96 hours of AMI in addition to the standard therapy.
  If there is no achievement of the target level of LDL-C, ≤1.5 mmol / L after 5-6 weeks from the AMI onset, patients additionally receive ezetimibe at a dose of 10 mg 1 time / day.
  Interventions: Drug: Atorvastatin 80mg
- Atorvastatin-Ezetimibe (Active Comparator): In the absence of reaching the target level of LDL-C of ≤1.4 mmol / L and a decrease in the indicator by ≥50% after 5-6 weeks from the onset of AMI, patients additionally receive ezetimibe at a dose of 10 mg 1 time / day.
  Interventions: Drug: Atorvastatin 80mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — Atorvastatin is prescribed at a dose of 80 mg / day from the first 24-96 hours of AMI in addition to the standard therapy
  Other Names: Ezetimibe

SUMMARY:
In a single-center, open-label, prospective, controlled, clinical study, it is planned to include 300 patients hospitalized in the cardiology department of SBHI Penza regional clinical hospital n.a. N.N. Burdenko. Recruitment of patients will be carried out at the Department of Therapy of the Medical Institute of the Penza State University. Patients meeting the inclusion criteria and not meeting the exclusion criteria will be included in the study.

Initially, lipid-lowering treatment with atorvastatin is prescribed at a dose of 80 mg / day from the first 24-96 hours of AMI in addition to the standard therapy.

If there is no achievement of the target level of LDL-C, ≤1.5 mmol / L after 5-6 weeks from the AMI onset, patients additionally receive ezetimibe at a dose of 10 mg 1 time / day.

Standard AMI treatment includes dual antiplatelet therapy, ACE inhibitors, beta-blockers (if indicated). Prescription of proton pump inhibitors and nitrates is possible (if indicated).

The total follow-up is 96 weeks. Prescreening - 600 people; screening and randomization - 300 people. Parameters of electrical myocardial heterogeneity, myocardial deformation characteristics, vascular rigidity, and quality of life will be assessed according to the study plan.

DETAILED DESCRIPTION:
Methods

1. Blood chemistry test. Total cholesterol, LDL, HDL, triglycerides, AST, ALT, CPK, glucose, CRP, creatinine, glycosylated hemoglobin
2. 2D and 3D transthoracic echocardiography (Vivid GE 95 Healthcare (USA). 3D speckle echocardiography (3DSTE) for a detailed study of the phase-by-phase movement and spatial interaction of all muscle layers of the left ventricle in different phases of the cardiac cycle to obtain quantitative values of the deformation of the left ventricle individual segments in the longitudinal, circumferential and radial directions.

   The analysis of standard indicators of echocardiography: biplane ejection fraction according to the Simpson method, 3D ejection fraction, EDV (end-diastolic volume), ESV (end-systolic volume) and their indices. The left ventricular myocardial mass index (LVMI).

   Using a tissue doppler, the parameters characterizing the diastolic function are recorded: the LA volume, the early diastolic velocity of the mitral valve fibrous ring, the ratio of the early diastolic transmitral flow E to the average early diastolic speed of the fibrous ring e´, and the maximum tricuspid regurgitation rate.

   Myocardial strain is analyzed using specialized software - EchoPac Software Only (General Electric Co., 2018). For three-dimensional strain analysis, the left ventricle is automatically divided into 17 segments using standard segmentation schemes. The software allows obtaining strain values in the endocardial, middle and epicardial layers of the myocardium. Over a period of time, indicators for each segment are automatically calculated:

   longitudinal strain/strain rate (LS,%/LSR, cm / s-1), circumferential strain/strain rate (CS,%/CSR, cm / s-1), radial strain/strain rate(RS,%/RSR, cm / s-1), area strain), rotation, rotation along the axis of the left ventricle (Torsion).
3. Long-term ECG monitoring over 3 leads with an assessment of the parameters of myocardial electrical instability A long-term ECG recording (120 hours) in patients with myocardial infarction will be performed using the Astrocard ECG system (CJSC Meditek, Russia) with 3-channel recorders. Long-term recordings will be analyzed separately for 3 time intervals: 24, 72 and 120 hours.

   Pauses of rhythm, rhythm disturbances - extrasystole, unstable tachycardia, AF paroxysm and atrial flutter, ventricular fibrillation, conduction disturbance will be recorded.

   Assessment of the ST segment dynamics will be carried out with detection of ischemia episodes, which will be detected when the ST segment is displaced ≥10 mV from the baseline 80 ms after the J point for at least 1 min - episodes of elevation and depression of the ST segment.

   According to the long-term ECG monitoring recordings, the following parameters will be analyzed (separately for 3 intervals - 24, 72 and 120 hours):

   circadian dynamics of heart rate; late ventricular potentials (LVP); variance and duration of the QT interval; heart rate variability (HRV); heart rate turbulence (TCP); chronotropic load (CL). Circadian dynamics of heart rate. The circadian dynamics of heart rate will be analyzed with an estimate of the minimum, average and maximum heart rate per day, during waking hours and night sleep. The circadian index (CI) will be defined as the ratio of the average heart rate in the daytime and the average heart rate in the night.

   LVP. The LVP will be evaluated in the standard averaging mode in the range of 40-100 Hz by the noise level not exceeding 0.9 μV. Records of the 24-h ECG in patients who have a decrease in intraventricular conduction, bundle branches blockade, will not be subjected to LVP analysis. An automatic analysis of late post-depolarization begins with a search for the QRS reference complex, which will be used later as a reference for averaging. Subsequently, the ECG signal will be processed programmatically by the time analysis method, at the end of which the following parameters will be evaluated: the width of the filtered QRS complex (QRSf), the duration of the low-amplitude potentials at the end of the QRS complex of the final part of the complex (HFLA), the rms value of the last 40 ms QRS (RMS ) Dispersion and QT interval duration. For a detailed study of the repolarization process in the analysis of records, close attention will be paid to the analysis of the duration, variability and variance of the QT interval.

   HRV. The following HRV time indicators will be considered:
   * Mean NN (ms) - average value of all RR-intervals;
   * SDNN (ms) - standard deviation of the average values of RR-intervals;
   * SDNNi (ms) - average value of standard deviations RR for 5-minute recording periods;
   * SDANN (ms) is the standard deviation of the mean values of the sinus intervals RR for 5 min;
   * rMSSD (ms) is the square root of the sum of the differences of subsequent RR intervals;
   * pNN50 (%) is the percentage of successive RR intervals differing by more than 50 ms;
   * HRVti - triangular index;
   * TINN is the index of triangular interpolation of the histogram of RR-intervals.

   HRV frequency parameters:
   * TotP (ms2) is the power of the total spectrum;
   * ULfP (ms2) - spectrum power in the ultralow frequency range;
   * VLfP (ms2) is the power of the spectrum within very low frequencies;
   * LfP (ms2) - low-frequency range of frequencies; HfP (ms2) - high-frequency component of HRV; L / H - an indicator of the balance of the vagosympathetic balance. Evaluation of the above HRV parameters will be carried out per day, night and day hours.

   TCP is characterized by two independent parameters - the beginning of turbulence (TO) and the slope of turbulence (TS).

   Heart CL is assessed by the level and duration of exceeding the actual (observed in the patient during monitoring) heart rate values of the threshold heart rate calculated individually according to the proposed formulas with differentiation for periods of wakefulness and night sleep:

   THR-W (bpm) = HRmax (bpm) × 0.45, where THR-W is the threshold value of the heart rate during wakeful hours in beats per minute, heart rate max is the age-appropriate value of the maximum possible heart rate in beats per minute, 0.45 is the coefficient of the threshold level of heart rate; THR-S (bpm) = THR-W (bpm): 1.24, where THR-S (bpm) is the threshold value of the heart rate during the night's sleep.
4. Ultrasound of the common carotid arteries with RF high frequency signal technology The study of local vascular stiffness by high-frequency RF signal technology using ultrasound of the common carotid arteries (CCA) will be carried out in B mode using MyLab 90 (Esaote, Italy).

   The RF signal technology includes two programs: RF-QIMT and RF-QAS. The following CCA indicators are analyzed: IMT - intima-media thickness, loc Psys - local systolic pressure in the carotid artery, loc Pdia - local diastolic pressure, P (T1) - pressure at the local point, stiffness indices β and α, DC is the coefficient of lateral distensibility, CC - coefficient of lateral compliance, Aix is the augmentation index, AP is the amplification pressure, PWV is the local pulse wave velocity in the carotid artery.
5. Ultrasound of the brachiocephalic and femoral arteries The brachiocephalic and femoral arteries will be scanned using a Vivid GE 95 ultrasound scanner (Healthcare, USA) using a linear sensor in B-mode, spectral Doppler imaging and color Doppler imaging.

   Quantitative analysis of atherosclerotic plaque includes determining the extent and degree of narrowing of the lumen of the vessel (percentage of stenosis) by the cross-sectional area (Sa) of the vessel:

   Sa = (A1 - A2) × 100% / A1, where A1 is the true cross-sectional area of the vessel, A2 is the passable cross-sectional area of the vessel.
6. Applanation tonometry. SphygmoCor apparatus (AtCor Medical, Australia) uses pulsed wave to calculate the characteristics of central pressure in aorta.

   The applanation tonometry technique includes two programs: PWA and PWV. The first allows to record central aortic pressure indicators: systolic aortic pressure - SBPao, diastolic - DBPao, pulse - PPao, mean hemodynamic - MBPao based on registration of the radial artery PWV. Using the PWV program, sequential recording of PWV from the common carotid and femoral arteries simultaneously with the ECG channel analyzes the PWV in the aorta (cfPWV).
7. Volume sphygmography. The measurements will be carried out with the VS-1000 device (Fukuda Denshi, Japan) while simultaneously recording plethysmograms on four limbs (using cuffs), ECG, phonocardiogram, and PWV on the carotid and femoral arteries.

   PWV is evaluated in different parts of the circulatory system (i.e., aorta (PWV), predominantly elastic arteries (R/L-PWV) and predominantly muscular arteries (B-PWV)).

   Cardio-Ankle Vascular Index (CAVI) is determined - an indicator that reflects the true stiffness of the vascular wall. CAVI is calculated by registering PWV at two points and measuring SBP and DBP. Additionally augmentation index and biological age will be calculated automatically.
8. Flow-mediated dilation. Endothelial function is evaluated by ultrasonic determination of flow-mediated dilation (FMD) during the postocclusive reactive hyperemia test using the method described by D. Celenmajer et. al.
9. Six-minute walk (6MW) test. The patient should not take cardiological drugs and should not smoke within at least 2 hours before the test. Before the 6MW test, the patient should have a 10-minute quiet rest in a sitting position. During this rest period, the following text should be read to the patient: "You will have to walk for 6 minutes, without using continuous running or alternate running and walking, with the aim to cover a maximum distance. You will walk back and forth along the corridor. You can slow down the pace, stop and have a rest in case of dyspnea or weakness. You can lean against the wall during rest. Then, you will have to resume the walk. Remember that your aim is to cover maximum distance in 6 minutes." At the 6-minute time point, the patient should be asked to stop and stand still until the covered distance has been measured.
10. Computer Pulse Oximetry. During the 6-minute walk test, computer pulse oximetry is planned on a PulseOx 7500 instrument (SPO medical, Israel) to study saturation dynamics in comparison groups.
11. Treatment compliance will be evaluated by standard methods (counting the remaining tablets). Morisky-Green Questionnaire
12. Quality of Life Assessment. The following questionnaires are planned to be completed: Seattle Angina Questionnaire (SAQ), Minnesota Questionnaire, Clinical Assessment Scale for CHF (MQCAS) (modified by Mareev VY, 2000), analog-visual scale.
13. Assessment of physical activity. It is planned to fill out a questionnaire for assessing the level of physical activity and a short international questionnaire for determining the physical activity of the International Questionnaire On Physical Activity - IPAQ
14. Assessment of Anxiety Depression. An analysis of anxiety and depressive disorders in patients using the hospital scale of anxiety and depression (HADS) is planned

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form 2 Primary STEMI or NSTEMI confirmed by ECG, troponin I and CPK-MB levels, coronary angiography.

3. Presence of an infarct-related artery according to coronary angiography.

Exclusion Criteria:

1. Presence of hemodynamically relevant stenosis exceeding 30% in several coronary arteries confirmed by CAG;
2. Recurrent or repeated myocardial infarction.
3. Exogenous hypertriglyceridemia (type 1 hyperchilomicronemia).
4. The development of acute heart failure III-IV prior to randomization
5. Individual intolerance to statins, ezetimibe.
6. Congenital and acquired heart diseases.
7. Severe concomitant diseases in the stage of decompensation.
8. Non-sinus rhythm, established artificial pacemaker.
9. Sinoatrial and atrioventricular blockade of 2-3 degrees.
10. QRS complex exceeding 100 ms.
11. The presence of severe LV hypertrophy according to echocardiography.
12. Uncontrolled hypertension with SBP> 180 mm Hg and DBP> 110 mmHg
13. Diabetes mellitus (DM) type 1 and 2.
14. Current existence of severe anemia (Hb < 100 g/L)
15. Chronic kidney disease (creatinine clearance less than 30 ml / min / 1.73 m2 according to the CKD-EPI).
16. Non-corrected thyroid dysfunction with hyper / hypothyroidism.
17. Body mass index (BMI) ≥35 kg / m2.
18. Pregnancy, lactation.
19. Alcohol abuse, drug addiction.
20. Other serious concomitant diseases that exclude the possibility of study participation.
21. Participation in other clinical trials within the last two months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2027-11-12 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias | up to 48 months
  Statistically significant differences in the frequency of ventricular arrhythmias as compared to controls
Systolic function | up to 48 months
  Statistically significant differences in systolic function of the left ventricle according to transthoracic echocardiography as compared to controls;
Myocardial deformation of the LA and LV | up to 48 months
  Statistically significant differences in the myocardial deformation of the LA and LV as compared to controls
PCI / CABG for a new case of coronary atherosclerosis, hospitalization for unstable angina | up to 48 months
  Statistically significant differences for major coronary events - PCI / CABG for a new case of coronary atherosclerosis, hospitalization for unstable angina as compared to controls
Myocardial electrical instability | up to 120 hours for 2 years period
  Statistically significant differences in the late ventricular potentials, heart rate variability, QT interval dispersion (ms) as compared to controls
Heart rate turbulence | up to 120 hours for 2 years period
  Statistically significant differences in the parameters of heart rate turbulence (%) as compared to controls

SECONDARY OUTCOMES:
Cardiovascular mortality | up to 48 months
  Statistically significant differences for incidence of CV events as compared to controls
Frequency of repeated fatal / non-fatal MI | up to 48 months
  Statistically significant differences in the frequency of repeated fatal / non-fatal MI as compared to controls
Hospitalization due to acute decompensation of heart failure | up to 48 months
  Statistically significant differences according to the frequency of hospitalization due to acute decompensation of heart failure as compared to controls
Structural state of arteries different types | up to 48 months
  Statistically significant differences in pulse wave velocities in arteries of various calibers, as compared to controls
Structural state of carotid artery | up to 48 months
  Statistically significant differences in intima-media thickness of carotid artery according ultrasound, as compared to controls
Functional state of arteries | up to 48 months
  Statistically significant differences in flow-mediated dilation parameters (diameter of brachial artery, mm) assessed by ultrasound, as compared to controls
Progression of CHF, exercise tolerance | up to 48 months
  Statistically significant differences in 6-minute walk test (distance covered, m), as compared to controls
Progression of CHF, laboratory data | up to 48 months
  Statistically significant differences in BNP level (pg/ml), as compared to controls
Left ventricular remodeling | up to 48 months
  Statistically significant differences echocardiographic parameters of left ventricle pathological remodeling (ejection fraction, %, EDVi, ESVi) as compared to controls
Lipid profile | up to 48 months
  Statistically significant differences of lipid profile (mmol/l) as compared to controls
Laboratory parameters | up to 48 months
  Statistically significant differences of CRP (mg/l) as compared to controls
Angina episodes | up to 48 months
  Statistically significant differences on angina episodes assessed by Seattle Angina Questionnaire (min - 19, max - 108 better outcome), as compared to controls
Quality of life questionnaire | up to 48 months
  Statistically significant differences according to the quality of life of patients assessed by Minnesota Questionnaire (min -0, max-105, worse outcome), as compared to controls
Quality of life questionnaire in СHF | up to 48 months
  Statistically significant differences according to the quality of life of patients assessed by Clinical Assessment Scale for CHF(min -0, max-20, worse outcome), as compared to controls
Patients wellbeing | up to 48 months
  Statistically significant differences of patients wellbeing according to the analog-visual scale , as compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Valentin E Oleynikov, DM, Principal Investigator — Penza State University
Locations (1):
- Valentin Oleynikov, Penza, Russia

IPD SHARING:
Plan to Share IPD: No